CLINICAL TRIAL: NCT02210559
Title: A Randomized, Open Label, Phase 1/2 Trial of Gemcitabine Plus Nab-paclitaxel With or Without FG-3019 as Neoadjuvant Chemotherapy in Locally Advanced, Unresectable Pancreatic Cancer
Brief Title: A Study of Gemcitabine Plus Nab-paclitaxel With or Without FG-3019 in Participants With Locally Advanced, Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-3019-069
Record Dates: First submitted 2014-07-31; First posted 2014-08-06 (Estimated); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer (Unresectable)
Keywords: locally; advanced; pancreatic; cancer; unresectable; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — pamrevlumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FG-3019 + Gemcitabine + Nab-paclitaxel (Experimental): Participants will receive FG-3019 35 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion on Days 1 and 15 of each treatment cycle and on Day 8 of the first cycle, gemcitabine 1000 mg/square meter (m^2) and nab-paclitaxel 125 mg/m^2 by IV infusion on Days 1, 8, and 15 of each treatment cycle. Treatment will be administered over a 28-day cycle, for up to 6 cycles.
  Interventions: Drug: FG-3019; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Gemcitabine + Nab-paclitaxel (Active Comparator): Participants will receive gemcitabine 1000 mg/ meter squared (m^2) and nab-paclitaxel 125 mg/m^2 by IV infusion on Days 1, 8, and 15 of each treatment cycle. Treatment will be administered over a 28-day cycle, for up to 6 cycles.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: FG-3019 — FG-3019 will be administered per dose and schedule specified in the arm group description.
  Arms: FG-3019 + Gemcitabine + Nab-paclitaxel
Drug: Gemcitabine — Gemcitabine will be administered per dose and schedule specified in the arm group description.
  Other Names: Gemzar
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered per dose and schedule specified in the arm group description.
  Other Names: Abraxane

SUMMARY:
This is a Phase 1/2 trial to evaluate the safety, tolerability, and efficacy of FG-3019 administered with gemcitabine and nab-paclitaxel in the treatment of locally advanced, unresectable pancreatic cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Male, or non-pregnant and, non-lactating female
* Histologically proven diagnosis of pancreatic ductal adenocarcinoma (PDAC)
* Radiographic and pathologic staging consistent with pancreatic cancer, locally advanced, unresectable (per National Comprehensive Cancer Network® [NCCN®] criteria)
* Laparoscopic confirmation that PDAC is locally advanced. Biliary stents are permitted.
* Measurable disease as defined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate liver, bone marrow, and renal function
* Agree to use contraception per protocol
* Less than Grade 2 pre-existing peripheral neuropathy

Key Exclusion Criteria:

* Prior chemotherapy or radiation for pancreatic cancer
* Solid tumor contact with superior mesenteric artery (SMA) >180°
* Previous (within the past 5 years) or concurrent malignancy diagnosis (expect non-melanoma skin cancer and in situ carcinomas)
* Major surgery, within 4 weeks prior to Day 1 on study
* History of allergy or hypersensitivity to human, humanized or chimeric monoclonal antibodies
* Exposure to another investigational drug within 42 days of first dosing visit, or 5 half-lives of the study product (whichever is longer)
* Uncontrolled intercurrent illness
* Any medical condition that, in the opinion of the Investigator, may pose a safety risk to a participant in this trial, may confound the assessment of safety and efficacy, or may interfere with study participation.
* Current abuse of alcohol or drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Picozzi, MD, Principal Investigator — Virginia Mason Medical Center - Benaroya Research Institute
Locations (8):
- United States (8):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Georgetown University - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center - Benaroya Research Institute, Seattle, Washington

REFERENCES:
- See also: Link to sponsor website where additional information is available regarding the investigational product and ongoing clinical trials. — http://www.fibrogen.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P): Participants received gemcitabine at 1000 milligrams (mg)/ meters (m)^2 plus nab-paclitaxel at 125 mg/m^2 by intraveneous (IV) infusion on Days 1, 8, and 15 of each cycle. Participants received pamrevlumab at 35 mg/kilograms (kg) by IV infusion on Days 1 and 15 of each cycle. An additional dose of pamrevlumab was given on Day 8 of the first cycle. Participants received a total of up to six 28-day cycles of treatment.
- Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP): Participants received gemcitabine at 1000 mg/ m^2 plus nab-paclitaxel at 125 mg/m^2 by IV infusion on Days 1, 8, and 15 of each cycle. Participants received a total of up to six 28-day cycles of treatment.
Period: Overall Study
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Started | 24 | 13
Received at Least 1 Dose of Study Drug | 24 | 13
Completed | 18 | 7
Not Completed | 6 | 6
Not completed — Progressive Disease | 3 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other than specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received any amount of study drugs including pamrevlumab, or gemcitabine, or nab-paclitaxel.
Groups:
- Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P): Participants received gemcitabine at 1000 mg/m^2 plus nab-paclitaxel at 125 mg/m^2 by IV infusion on Days 1, 8, and 15 of each cycle. Participants received pamrevlumab at 35 mg/kg by IV infusion on Days 1 and 15 of each cycle. An additional dose of pamrevlumab was given on Day 8 of the first cycle. Participants received a total of up to six 28-day cycles of treatment.
- Total: Total of all reporting groups
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP) | Total
Number analyzed (Participants) | 24 | 13 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (7.75) | 60.8 (9.18) | 64.4 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 13 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 22 | 10 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as a new or worsening AE that occurred in the window of first infusion of any study drug (Day 1) and within 28 days of the last infusion of study drug or the day before surgery, whichever occurred first. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: From first infusion of any study drug (Day 1) up to 28 days after last infusion of study drug or the day before surgery (up to Day 196)
Population: Safety population included all participants who had received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
Participants
  TEAEs | 24 | 12
  SAEs | 9 | 6

2. Primary Outcome: Number of Participants Who Had Surgical Complications Post-Resection
Description: Number of participants who had surgical complications (for example; surgical site infection, intra-abdominal abscess, or perioperative leak during surgery) has been reported
Time Frame: 30 days following discharge after surgery (up to Day 198)
Population: ITT population included all randomized participants who received any amount of study drugs including pamrevlumab, or gemcitabine, or nab-paclitaxel.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Became Eligible for Surgery
Time Frame: After completion of 24 weeks of treatment with study drug
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
Participants | 17 | 2

4. Secondary Outcome: Number of Participants in Whom R0 Resection Was Achieved
Description: R0 resection was determined by pathological examination of the surgical specimen after resection.
Time Frame: After completion of 24 weeks of treatment with study drug
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
Participants | 4 | 1

5. Secondary Outcome: Number of Participants in Whom R0 or R1 Resection Was Achieved
Description: R0 or R1 resection was determined by pathological examination of the surgical specimen after resection.
Time Frame: After completion of 24 weeks of treatment with study drug
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
Participants | 8 | 1

6. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR) Per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduced in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
Participants | 5 | 3

7. Secondary Outcome: Median Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: From randomization until death from any cause, assessed up to 4 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
months | 19.38 [13.34 to 27.73] | 23.47 [13.27 to 46.46]

8. Secondary Outcome: Median Progression-Free Survival
Description: Progression-free survival was defined as the time from randomization until objective tumor progression or death. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From randomization until objective tumor progression or death, assessed up to 4 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
Number analyzed (Participants) | 24 | 13
months | 14.11 [8.25 to 18.40] | 11.63 [3.88 to 20.40]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from first infusion of any study drug (Day 1) up to 28 days after last infusion of study drug or the day before surgery (up to Day 196). All-Cause Mortality was assessed from first infusion of any study drug until death, assessed up to 4 years.
Description: Safety population included all participants who had received any dose of study drug.
Arm/Group | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP)
All-Cause Mortality (participants affected / at risk) | 17/24 | 7/13
Serious Adverse Events (participants affected / at risk) | 9/24 | 6/13
Other Adverse Events (participants affected / at risk) | 24/24 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) (N=24) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP) (N=13)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopthy (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Device occlusions (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Gemcitabine Plus Nab-paclitaxel + Pamrevlumab (G/NP+P) (N=24) | Arm B: Gemcitabine Plus Nab-paclitaxel (G/NP) (N=13)
Neutropenia (Blood and lymphatic system disorders) | 9 | 4
Anaemia (Blood and lymphatic system disorders) | 9 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 3 | 0
Dry eye (Eye disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 17 | 7
Diarrhoea (Gastrointestinal disorders) | 12 | 7
Constipation (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 3 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 18 | 10
Oedema peripheral (General disorders) | 14 | 5
Pyrexia (General disorders) | 7 | 2
Chills (General disorders) | 5 | 1
Gait disturbance (General disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Cellulitis (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 0
Rash pustular (Infections and infestations) | 1 | 1
Body tinea (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 2
Platelet count decreased (Investigations) | 8 | 1
Alanine aminotransferase increased (Investigations) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 2
Blood alkaline phosphatase increased (Investigations) | 4 | 2
Weight decreased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 10 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 4
Dizziness (Nervous system disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 3 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Nocturia (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 7
Rash (Skin and subcutaneous tissue disorders) | 7 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02210559/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT02210559/SAP_001.pdf